CLINICAL TRIAL: NCT06592846
Title: FERtility After Therapy With Intensive Lymphoma in Young Women: LNH-03 1B, LNH-03 2B, LNH-07 3B, GAINED Follow-up
Acronym: FERTILE
Status: Completed | Type: Observational
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Other Study IDs: FERTILE
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-01

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The FERTILE study is a retrospective cohort study evaluating fertility after intensive treatment with RCHOP14/RCHOP21 or ACVBP in young patients with diffuse large B-cell lymphoma treated in clinical trials conducted by the LYSA group and still alive several years after the end of the trial.

DETAILED DESCRIPTION:
The FERTILE study is a retrospective cohort study evaluating fertility after intensive treatment with RCHOP14/RCHOP21 or ACVBP in young patients (≤ 38 years) with diffuse large B-cell lymphoma treated in 4 clinical trials conducted by the LYSA group and still alive several years after the end of the trial.

Chemotherapy treatments used to treat diffuse large B-cell lymphoma in women of childbearing age may cause loss of fertility.

There are few studies dedicated specifically to women treated for non-Hodgkin's lymphoma, particularly in the context of intensive CHOP-based regimens (R-CHOP14/R-CHOP21/R-ACVBP). These studies do not provide any details on the type of treatment and the clinical characteristics of the patients. It is in this context that we propose the FERTILE study.

This study is based on the collection and reuse of data already available in the LNH03-1B, LNH03-2B, LNH07-3B and GAINED clinical trials such as the age of the patients, the treatments, the diagnosis. The results of hormonal assessments and fertility tests (endovaginal ultrasound) will also be consulted in the medical file.

In addition, a questionnaire concerning fertility will be proposed by the physician-investigator.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects are women
2. Participation in one of the following clinical trials: LNH 03 1B or LNH 03 2B or LNH 07 3B or GAINED
3. Age at initial diagnosis between 18 years and 38 years inclusive, which has allowed their inclusion in the clinical trial
4. Treated with R-ACVBP or R-CHOP14/R-CHOP21 in these clinical trials
5. No relapse of their diffuse large B-cell lymphoma
6. Possible use of stem cell transplantation during clinical trials
7. Subjects are still alive today

Exclusion Criteria:

1. Subjects died
2. Subjects lost to follow-up

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The subjects are women
Study Population: Young patients ( ≤ 38 years of age) with diffuse large B-cell lymphoma treated with intensive RCHOP or ACVBP chemotherapy in clinical trials conducted by the LYSA group, and still alive several years after the end of the the trial
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Study fertility by evaluating the rate of spontaneous pregnancy (with live-born children) in women (≤ 38 years) treated for diffuse large B-cell lymphoma in 4 LYSA clinical trials. | Day 0 from date of questionnaire signature
  The fertility rate: spontaneous pregnancy rate (with live births) among young women who wish to have children.

SECONDARY OUTCOMES:
Identify the predictive factors associated with pregnancy success after intensive chemotherapy treatment. | Day 0 from date of questionnaire signature
  Identification of predictive factors associated with pregnancy after lymphoma treatment, assessed by a Cox proportional hazards model.
Identify predictive factors associated with gonadal dysfunction. | Day 0 from the questionnaire signature
  The identification of predictive factors associated with gonadal dysfunction after lymphoma treatment, assessed by a Cox proportional hazards model.
  Methods used to assess ovarian reserve (biochemical tests including basal levels of including basal levels of FSH, LH, estradiol and antimüllerian hormone; ultrasound estradiol and antimüllerian hormone; ultrasound measurements including number of antral follicles and ovarian volume).
Study the different clinical practices concerning the preservation of fertility in LYSA sites. | Day 0 from date of questionnaire signature
  Fertility preservation techniques used in the centres (ovarian stimulation, cryopreservation of ovarian tissue, GnRH agonists, in vitro maturation).
  Methods used to assess ovarian reserve (biochemical tests including basal levels of including basal levels of FSH, LH, estradiol and antimüllerian hormone; ultrasound estradiol and antimüllerian hormone; ultrasound measurements including number of antral follicles and ovarian volume)

CONTACTS AND LOCATIONS:
Overall Officials: Lucie OBERIC, MD, Principal Investigator — Institut Universitaire du Cancer Toulouse - Oncopole
Locations (27):
- France (27):
  - CH d'Avignon - Hôpital Henri Duffaut, Avignon
  - Institut d'Hématologie de Basse Normandie (IHBN), Caen
  - APHP - Hôpital Henri Mondor, Créteil
  - CHU de Dijon - Hôpital François Mitterand, Dijon
  - CHD de Vendée, La Roche-sur-Yon
  - Groupe Hospitalier La Rochelle-Ré-Aunis, La Rochelle
  - CHU de Grenoble - Hôpital Albert Michallon, La Tronche
  - CH de Versailles - Hôpital André Mignot, Le Chesnay
  - CH St Vincent de Paul, Lille
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - CHU de Limoges - Hôpital Universitaire Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU d'Orléans, Orléans
  - APHP - Hôpital Saint Louis, Paris
  - APHP - Hôpital de la Pitié Salpétrière, Paris
  - APHP - Hôpital Necker, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Poitiers - Hôpital de la Milétrie, Poitiers
  - CH Annecy Genevois, Pringy
  - CHU de Reims - Hôpital Robert Debré, Reims
  - Centre Henri Becquerel, Rouen
  - CHU de Saint Etienne_I.CHU.SE, Saint-Priest-en-Jarez
  - IUCT Oncopole de Toulouse, Toulouse
  - CHU de Nancy - Hôpital de Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ketterer N, Coiffier B, Thieblemont C, Ferme C, Briere J, Casasnovas O, Bologna S, Christian B, Connerotte T, Recher C, Bordessoule D, Fruchart C, Delarue R, Bonnet C, Morschhauser F, Anglaret B, Soussain C, Fabiani B, Tilly H, Haioun C. Phase III study of ACVBP versus ACVBP plus rituximab for patients with localized low-risk diffuse large B-cell lymphoma (LNH03-1B). Ann Oncol. 2013 Apr;24(4):1032-7. doi: 10.1093/annonc/mds600. Epub 2012 Dec 12. PMID 23235801
- [Background] Recher C, Coiffier B, Haioun C, Molina TJ, Ferme C, Casasnovas O, Thieblemont C, Bosly A, Laurent G, Morschhauser F, Ghesquieres H, Jardin F, Bologna S, Fruchart C, Corront B, Gabarre J, Bonnet C, Janvier M, Canioni D, Jais JP, Salles G, Tilly H; Groupe d'Etude des Lymphomes de l'Adulte. Intensified chemotherapy with ACVBP plus rituximab versus standard CHOP plus rituximab for the treatment of diffuse large B-cell lymphoma (LNH03-2B): an open-label randomised phase 3 trial. Lancet. 2011 Nov 26;378(9806):1858-67. doi: 10.1016/S0140-6736(11)61040-4. PMID 22118442
- [Background] Casasnovas RO, Ysebaert L, Thieblemont C, Bachy E, Feugier P, Delmer A, Tricot S, Gabarre J, Andre M, Fruchart C, Mounier N, Delarue R, Meignan M, Berriolo-Riedinger A, Bardet S, Emile JF, Jais JP, Haioun C, Tilly H, Morschhauser F. FDG-PET-driven consolidation strategy in diffuse large B-cell lymphoma: final results of a randomized phase 2 study. Blood. 2017 Sep 14;130(11):1315-1326. doi: 10.1182/blood-2017-02-766691. Epub 2017 Jul 12. PMID 28701367
- [Background] Le Gouill S, Ghesquieres H, Oberic L, Morschhauser F, Tilly H, Ribrag V, Lamy T, Thieblemont C, Maisonneuve H, Gressin R, Bouhabdallah K, Haioun C, Damaj G, Fornecker L, Bouhabdallah R, Feugier P, Sibon D, Cartron G, Bonnet C, Andre M, Chartier L, Ruminy P, Kraeber-Bodere F, Bodet-Milin C, Berriolo-Riedinger A, Briere J, Jais JP, Molina TJ, Itti E, Casasnovas RO. Obinutuzumab vs rituximab for advanced DLBCL: a PET-guided and randomized phase 3 study by LYSA. Blood. 2021 Apr 29;137(17):2307-2320. doi: 10.1182/blood.2020008750. PMID 33211799